CLINICAL TRIAL: NCT05420987
Title: The Effects of JING SI HERBAL TEA LIQ UID PACKETS on Inflammation in Patients With Cardiovascular Disease
Brief Title: Effect of Jing Si Herbal Tea on Inflammation in Patients With Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB111-025-A
Record Dates: First submitted 2022-05-29; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Response; Gut Microbiome; Life Quality; Trimethylamine N-oxide; Cardiovascular Diseases; Herbal Medicine
Keywords: Jing Si herbal tea liquid packet; microbiome; trimethylamine N-oxide (TMAO); double-blind randomized controlled trial
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active arm (Experimental): Jing Si herbal tea liquid packet
  Interventions: Dietary Supplement: Jing Si herbal tea liquid packet
- control arm (Placebo Comparator): Jing Si herbal tea placebo
  Interventions: Dietary Supplement: Jing Si herbal tea liquid packet

INTERVENTIONS:
Dietary Supplement: Jing Si herbal tea liquid packet — Jing Si herbal tea includes eight Taiwan native-grown herbs: such as mugwort leaves, fish needle grass, Ophiopogon japonicus, platycodon, perilla leaves, chrysanthemum, and licorice

SUMMARY:
Jing Si herbal tea includes eight Chinese herbs: such as mugwort leaves, fish needle grass, Ophiopogon japonicus, platycodon, perilla leaves, chrysanthemum, and licorice. In vitro, these ingredients were found to be able to block the binding of SARS-CoV-2 and human ACE2 receptor, and further reduce the penetration ability of the virus. Now, Jing Si herbal tea liquid packets have obtained the special license for export from the Ministry of Health and Welfare in Taiwan.

The aim of the study is to investigate (1) the effect of Jing Si herbal tea liquid on blood pressure, blood sugar, and cholesterol in patients with cardiovascular diseases. (2)The human gut microbiota change which is associated with TMAO production (3) The proinflammatory and inflammatory biomarkers change.

We are going to recruit 100 participants from cardiovascular clinics, including patients with hypertension, hyperlipidemia, ischemic heart disease and diabetes, aged 20-75 years old. We exclude those who are cancer patients, have comorbidities with poor control, patients with eGFR< 40 ml/min/1.73m2, those who are pregnant, breastfeeding, and in their menstrual period when recruiting.

The study has two parts. The first part is a pilot study with 20 subjects all take active Jing Si herbal tea. The second part is a double-blind randomized controlled study with 40 subjects in each arm.

DETAILED DESCRIPTION:
Jing Si herbal tea includes eight Chinese herbs: such as mugwort leaves, fish needle grass, Ophiopogon japonicus, platycodon, perilla leaves, chrysanthemum, and licorice. In vitro, these ingredients were found to be able to block the binding of SARS-CoV-2 and human ACE2 receptor, and further reduce the penetration ability of the virus. Now, Jing Si herbal tea liquid packets have obtained the special license for export from the Ministry of Health and Welfare in Taiwan.

The aim of the study is to investigate (1) the effect of Jing Si herbal tea liquid on blood pressure, blood sugar, and cholesterol in patients with cardiovascular diseases. (2)The human gut microbiota change which is associated with TMAO production (3) The proinflammatory and inflammatory biomarkers change.

We are going to recruit 100 participants from cardiovascular clinics, including patients with hypertension, hyperlipidemia, ischemic heart disease and diabetes, aged 20-75 years old. We exclude those who are cancer patients, have comorbidities with poor control, patients with eGFR< 40 ml/min/1.73m2, those who are pregnant, breastfeeding, and in their menstrual period when recruiting.

The study has two parts. The first part is a pilot study with 20 subjects all take active Jing Si herbal tea. The second part is a double-blind randomized controlled study with 40 subjects in each arm.

All the patients' specimens and questionnaires are going to be collected on Day0, Day28, and Day84.

ELIGIBILITY:
Inclusion Criteria:

* hypertension,
* hyperlipidemia,
* ischemic heart disease
* diabetes

Exclusion Criteria:

* cancer patients,
* have comorbidities with poor control
* patients with eGFR< 40 ml/min/1.73m2
* who are pregnant, breastfeeding, and in their menstrual period when recruiting

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
inflammatory biomarkers | 3 months
  IL-1b (pg/mL), IL-4(pg/mL), IL-6(pg/mL), IL-10(pg/mL), TNF-gamma(pg/mL),TNF-alpha (pg/mL)
inflammatory biomarkers | 3 months
  GlycA (umol/L)
lipid profile , Glu-AC, hs_CRP | 3 months
  Total cholesterol(mg/dL), TG(mg/dL), HDL-C(mg/dL), LDL-C(mg/dL), uric acid (mg/dL) and Glu-AC (mg/dL),hs_CRP(mg/dL)
diabetes control index | 3 months
  HbA1c (%), insulin (mU/L), HOMA-IR, HOMA-beta
biomarkers for congestive heart failure | 3 months
  Nt-proBNP (pg/ mL)
heart function measurement for congestive heart failure | 3 months
  LVEF(%)
kidney function 1 | 3 months
  BUN (mg/dL),Cre (mg/dL)
kidney function 2 | 3 months
  eGFR (mL/min)
kidney function 3 | 3 months
  Urine Albumin to Creatinine Ratio(mg/g)
Gut microbiome | 3 months
  TMAO (uM)
immune composition analysis 1 | 3 months
  CD3(%), CD4(%), CD8(%), CD56(%), CD11b(%), Foxp3(%), NK,HLA-DR(%)
immune composition analysis 2 | 3 months
  WBC (10^3/uL)
immune function analysis | 3 months
  IFN-gamma (IU/mL)

IPD SHARING:
Plan to Share IPD: No
no, we are not going to share IPD.